CLINICAL TRIAL: NCT04452006
Title: Single-center, Double-blind, Randomized, Placebo-controlled, Three-part, First-in-human, Phase 1 Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of ACT-541478 in Healthy Subjects
Brief Title: A Study in Healthy Subjects to Investigate the Safety and Tolerability of ACT- 541478 as Well as What ACT-541478 Does to the Body and the Way the Body Takes up, Distributes, and Gets Rid of ACT-541478
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Based on interim analysis, the Sponsor decided to terminate the study prematurely.
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: ID-088-101
Record Dates: First submitted 2020-06-26; First posted 2020-06-30 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-07

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Part A: Single-ascending dose study in healthy male subjects (including investigation of the effect of food); Part B: Single-dose, three-way crossover study in healthy male subjects to investigate specific/additional parameters related to safety and tolerability; Part C: Multiple-ascending dose study in healthy male and female subjects (including healthy male and female elderly subjects).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (11):
- Part A (SAD) - A1, ACT-541478 10 mg fasted (Experimental): SAD = single ascending dose
  Interventions: Drug: ACT-541478 10 mg; Drug: Matching placebo
- Part A (SAD) - A2, ACT-541478 30 mg fasted (Experimental): SAD = single ascending dose
  Interventions: Drug: ACT-541478 30 mg; Drug: Matching placebo
- Part A (SAD) - A3 (Period 1), ACT-541478 100 mg fasted (Experimental): SAD = single ascending dose
  Interventions: Drug: ACT-541478 100 mg; Drug: Matching placebo
- Part A (SAD) - A3 (Period 2), ACT-541478 100 mg fed (Experimental): SAD = single ascending dose
  Interventions: Drug: ACT-541478 100 mg; Drug: Matching placebo
- Part A (SAD) - A4, ACT-541478 300 mg fasted (Experimental): SAD = single ascending dose
  Interventions: Drug: ACT-541478 300 mg; Drug: Matching placebo
- Part A (SAD) - A5, ACT-541478 1000 mg fasted (Experimental): SAD = single ascending dose
  Interventions: Drug: ACT-541478 1000 mg; Drug: Matching placebo
- Part B - B1-3, ACT-541478 low or high dose (Experimental)
  Interventions: Drug: ACT-541478 high or low dose (or placebo); Drug: Matching placebo
- Part C (MAD) - C1, ACT-541478 30 mg, fasted (Experimental): MAD = multiple ascending dose
  Interventions: Drug: ACT-541478 30 mg; Drug: Matching placebo
- Part C (MAD) - C2, ACT-541478 100 mg, fasted (Experimental): MAD = multiple ascending dose
  Interventions: Drug: ACT-541478 100 mg; Drug: Matching placebo
- Part C (MAD) - C3, ACT-541478 300 mg, fasted (Experimental): MAD = multiple ascending dose
  Interventions: Drug: ACT-541478 300 mg; Drug: Matching placebo
- Part C (Elderly) E1, ACT-541478, fasted (Experimental)
  Interventions: Drug: ACT-541478 dose E1; Drug: Matching placebo

INTERVENTIONS:
Drug: ACT-541478 10 mg — ACT-541478 will be provided in HPMC capsules for oral administration at a dose strength of 10 mg.
  Arms: Part A (SAD) - A1, ACT-541478 10 mg fasted
Drug: ACT-541478 30 mg — ACT-541478 will be provided in HPMC capsules for oral administration at a dose strength of 10 mg.
  Arms: Part A (SAD) - A2, ACT-541478 30 mg fasted; Part C (MAD) - C1, ACT-541478 30 mg, fasted
Drug: ACT-541478 100 mg — ACT-541478 will be provided in HPMC capsules for oral administration at a dose strength of 50 mg.
  Arms: Part A (SAD) - A3 (Period 1), ACT-541478 100 mg fasted; Part A (SAD) - A3 (Period 2), ACT-541478 100 mg fed; Part C (MAD) - C2, ACT-541478 100 mg, fasted
Drug: ACT-541478 300 mg — ACT-541478 will be provided in HPMC capsules for oral administration at dose strengths of 50 mg and 250 mg.
  Arms: Part A (SAD) - A4, ACT-541478 300 mg fasted; Part C (MAD) - C3, ACT-541478 300 mg, fasted
Drug: ACT-541478 1000 mg — ACT-541478 will be provided in HPMC capsules for oral administration at a dose strength of 250 mg.
  Arms: Part A (SAD) - A5, ACT-541478 1000 mg fasted
Drug: ACT-541478 high or low dose (or placebo) — Cross-over design: ACT-541478 will be provided in HPMC capsules for oral administration at high or low dose strengths (to be defined after completion of Part A).
  Arms: Part B - B1-3, ACT-541478 low or high dose
Drug: ACT-541478 dose E1 — E1 is a dose level that has been investigated and well tolerated in the adult dose level groups C1 to C3. ACT-541478 will be provided in HPMC capsules for oral administration at dose strengths of 10, 50, and 250 mg.
  Arms: Part C (Elderly) E1, ACT-541478, fasted
Drug: Matching placebo — Matching placebo will be provided in HPMC capsules for oral administration.

SUMMARY:
A study in healthy subjects to investigate the safety and tolerability of ACT-541478 as well as what ACT-541478 does to the body and the way the body takes up, distributes, and gets rid of of ACT-541478

ELIGIBILITY:
Inclusion Criteria:

Part A/B/C:

* Signed informed consent in a language understandable to the subject prior to any study-mandated procedure.
* BMI of 18.0 to 29.9 kg/m2 (inclusive) at Screening.
* SBP 100-139 mmHg, DBP 50-89 mmHg, and pulse rate 50-90 bpm (inclusive), measured on either arm, after 5 min in the supine position at Screening and on Day -1 in the first period, if applicable.
* Fertile male subjects (defined as physiologically capable of conceiving a child according to the investigator's judgment) must agree to refrain from fathering a child and:

  1. be sexually abstinent with women of child-bearing potential or use condoms during sexual intercourse with women of child-bearing potential from (first) study treatment administration up to at least 90 days after (last) study treatment administration. Moreover, it is recommended that women of child-bearing potential partners of male subjects consistently and correctly use for the same period a highly effective method of contraception with a failure rate of < 1% per year.
  2. to not donate sperm from (first) study treatment administration up to at least 90 days after (last) study treatment administration.
* Body temperature in the range of 35.5° to 37.5 °C at Screening and on Day -1 in the first period, if applicable.
* 12-lead safety ECG: QTcF ≤ 450 ms, QRS ≤ 110 ms, PR ≤ 220 ms, and resting HR 50-90 bpm (inclusive) with no clinically relevant abnormalities on 12-lead safety ECG after at least 5 min in the supine position at Screening and on Day -1 in the first period, if applicable.
* Normal renal function as confirmed by an estimated glomerular filtration rate ≥ 80 mL/min/1.73 m2 determined at Screening using the Chronic Kidney Disease Epidemiology Collaboration formula.

Part A/B:

- Healthy male subjects aged between 18 and 55 years (inclusive) at Screening.

Parts C1 to C3 (Adult subjects):

- Healthy male and female subjects aged between 18 and 55 years (inclusive) at Screening.

Parts E1 and E2 (Elderly subjects):

- Healthy male and female subjects aged between 65 and 80 years (inclusive) at Screening.

Parts C1 to C3, E1 and E2 (Female subjects):

* Women of child-bearing potential must have a negative serum pregnancy test at Screening and a negative urine pregnancy test on Day
* 1. They must consistently and correctly use (from Screening, during the entire study, and for at least 30 days after last study treatment administration) a highly effective method of contraception with a failure rate of < 1% per year, or be sexually inactive, or have a vasectomized partner. If a hormonal contraceptive is used, it must have been initiated at least 1 month before first study treatment administration.
* Women of child-bearing potential (i.e., postmenopausal [defined as 12 consecutive months with no menses without an alternative medical cause, confirmed by an FSH test > 40 mIU/mL], or with documented previous bilateral salpingectomy, bilateral salpingo oophorectomy or hysterectomy, or with premature ovarian failure [confirmed by a specialist], XY genotype, Turner syndrome, uterine agenesis).

Exclusion Criteria:

Part A/B/C

* History of major medical or surgical disorders, which, in the opinion of the investigator, are likely to interfere with the absorption, distribution, metabolism, or excretion of the study treatment (appendectomy and herniotomy allowed, cholecystectomy not allowed).
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol.
* History or presence of cardiac rhythm disorders (e.g., sinoatrial heart block, sick-sinus syndrome, 2nd or 3rd degree AV block, long QT syndrome, symptomatic bradycardia, atrial flutter, or atrial fibrillation).
* Any illness with a potential to increase the risk of the subject based on medical history.
* Clinically relevant findings in clinical laboratory tests (hematology, clinical chemistry, and urinalysis) at Screening (and on Day -1 in Part A and C) or any of the following laboratory parameters out of normal range: ALT, AST, total bilirubin, creatinine, TSH, and/or hemoglobin, at Screening and on Day -1 in the first period, if applicable.
* Any signs or symptoms of active, ongoing infection judged to be clinically relevant by the investigator (special attention should be given to clinical signs and symptoms consistent with COVID-19).

Part A (A3, effect of food)

* Known lactose intolerance.
* Known hereditary problems of galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption.
* Inability or unwillingness to completely consume the required high-fat meal.

Part C

* Pregnant or lactating women.
* Relevant history of a suicide attempt or suicidal behavior. Any recent suicidal ideation within the last 6 months (categories 4 or 5), or any suicidal behavior within the last 2 years, except for "Non-Suicidal Self-Injurious Behavior" (item also included in the Suicidal Behavior section), as judged by the investigator using the Columbia-Suicide Severity Rating Scale (C-SSRS) at Screening.
* Result ≤ 27 in the Mini-Mental State Examination (MMSE®2™), assessed at Screening (E1 and E2 only).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2021-04-20 (Actual); Study Completion 2021-04-20 (Actual)

PRIMARY OUTCOMES:
Treatment-emergent (serious) AEs | From (first) study treatment administration up to 96 h after last study treatment administration in the corresponding period (if applicable). Total duration: up to 5 days.

OTHER OUTCOMES:
Plasma PK parameters of ACT-541478 - Part A and B, incl. A3 (fed condition): Cmax | Blood samples for PK analysis will be taken at various timepoints. Total duration: up to 5 days.
Plasma PK parameters of ACT-541478 - Part A and B, incl. A3 (fed condition): tmax | Blood samples for PK analysis will be taken at various timepoints. Total duration: up to 5 days.
Plasma PK parameters of ACT-541478 - Part A and B, incl. A3 (fed condition): AUC0-inf | Blood samples for PK analysis will be taken at various timepoints. Total duration: up to 5 days.
Plasma PK parameters of ACT-541478 - Part A and B, incl. A3 (fed condition): t½ | Blood samples for PK analysis will be taken at various timepoints. Total duration: up to 5 days.
Plasma PK parameters of ACT-541478 - Part C, incl. C1 to C3 (adults) and E1 (elderly): Cmax | Blood samples for PK analysis will be taken at various timepoints. Total duration: up to 5 days.
Plasma PK parameters of ACT-541478 - Part C, incl. C1 to C3 (adults) and E1 (elderly): tmax | Blood samples for PK analysis will be taken at various timepoints. Total duration: up to 5 days.
Plasma PK parameters of ACT-541478 - Part C, incl. C1 to C3 (adults) and E1 (elderly): AUCτ | Blood samples for PK analysis will be taken at various timepoints. Total duration: up to 5 days.
Plasma PK parameters of ACT-541478 - Part C, incl. C1 to C3 (adults) and E1 (elderly): t1/2 | Blood samples for PK analysis will be taken at various timepoints. Total duration: up to 5 days.
Specific/additional parameters related to safety and tolerability - Part B | At various timepoints. Total duration: up to 5 days.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Idorsia Pharmaceuticals Ltd.
Locations (1):
- Parexel International GmbH, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No